CLINICAL TRIAL: NCT06700005
Title: ReadMap: Reading in Stroke Alexia and Typical Aging
Acronym: ReadMap
Status: Recruiting | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: MedStar National Rehabilitation Network (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ReadMap; R01DC020446 (NIH)
Record Dates: First submitted 2024-11-06; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Aphasia; Stroke; Alexia
Keywords: aphasia; stroke; brain injury; speech; language; reading; alexia; apraxia
MeSH Terms: conditions — Aphasia; Stroke; Dyslexia; Brain Injuries; Speech; Language; Apraxias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Survivors: Participants have had a left-hemisphere stroke, or a stroke elsewhere in the brain causing aphasia or alexia (i.e., reading difficulties). They are given a series of standardized and in-house tests of reading, language and cognition to provide a detailed profile of strengths and weaknesses, plus an MRI.
- Controls: Participants are matched to the stroke cohort in age, educational background, race, and gender but have no history of brain injury. They are also given a series of standardized and in-house tests of reading, language and cognition to provide a detailed profile of strengths and weaknesses, plus an MRI.

SUMMARY:
Loss of reading ability due to stroke, called alexia, likely affects over a million Americans at any given time and causes difficulty performing many daily life functions, such as paying bills, using email/text, reading for pleasure, and reading signs in the community. Understanding the brain and cognitive basis of alexia could improve diagnosis and treatment of this important problem. In this study, the investigators will perform a large-scale behavioral and brain imaging study of stroke survivors and typical older adults to improve our understanding of the brain and cognitive basis of reading in both of these groups.

Participants will complete a battery of tests of reading, speech, language, and thinking abilities. In addition, some participants will complete an MRI. Sessions will be completed across approximately 2-6 weeks, but may be extended depending on participants' schedules and availability. Some participants will be invited to repeat these procedures once or twice in approximately 3-12 months to monitor for changes in reading abilities and MRI measurements over time.

ELIGIBILITY:
Inclusion criteria:

Stroke Survivors:

* Age >= 18
* Learned English at 8 years or younger
* Brain injury resulting from stroke

Controls:

* Age >= 18
* Learned English at 8 years or younger

Exclusion criteria for all groups:

* History of other brain disorder that could interfere with our ability to interpret results (e.g., Multiple sclerosis, dementia, head injury causing loss of consciousness)
* Severe psychiatric condition that would interfere with participation in the study
* History of diagnosed learning disorder
* Hearing or vision loss that interferes with performance on behavioral tests even after correction with glasses/hearing aids.
* Inability to follow study procedures despite maximal support

Additional exclusion criteria for MRIs:

* Presence of metal in the body that is incompatible with MRI
* Pregnancy
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are survivors of left hemisphere stroke with or without reading difficulties, or people with aphasia or alexia due to strokes in other parts of the brain. The investigators recruit participants primarily from the Washington, DC region, but some participants may travel from farther away to participate in the study. The investigators aim for our participants to be fully representative of the diversity of individuals with stroke in the general population.
  Control participants have not had a stroke or other brain injury, and are matched to stroke survivors on age, gender, race, educational background, and stroke risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
MP-RAGE (Magnetization Prepared Rapid Acquisition Gradient Echo) | Collected within 1 month of behavioral testing
  Part of MRI sequence that measures deep grey matter structure.
DTI (Diffusion Tensor Imaging) | Collected within 1 month of behavioral testing
  Part of MRI sequence that measures the rate of water diffusion between cells to understand and create a map of internal structures.
Behavioral testing | Collected within 1 month of MRI
  Battery of standard clinical and in-house behavioral tests to measure speech, language, and cognition. Final score is derived from principle components analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Turkeltaub, MD,PhD, Principal Investigator — Georgetown University; MedStar National Rehabilitation Hospital
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States